CLINICAL TRIAL: NCT04200014
Title: Bradycardia High Risk Patient Identification After Syncope With Loop Recorder an Observational Study in Nancy University Hospital
Brief Title: Bradycardia Risk Stratification With Loop Recorder After Syncope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI198
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Implantable Loop Recorder
Keywords: Syncope; Arrhythmia
MeSH Terms: conditions — Syncope; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Syncope and Implantable loop recorder: Patients implanted with a subcutaneous Loop Recorder after syncope in Nancy University Hospital

SUMMARY:
Syncope is a common symptom that may be related to a conductive disorder. If no bradycardia is authenticated, it is often necessary to implant an implantable loop recorder.

In somes cases, implantable loop recorder records cardiac conductive disorders. In this study, we want to try to identify a group of patients for whom we could immediately implant a pacemaker without prior implantation of an implantable loop recorder given the high probability of implantation of a pacemaker after interrogation of the implantable loop recorder. It would be interesting for the reduction of interventions for the patients and for the economic aspect of the healthcare system

ELIGIBILITY:
Inclusion Criteria:

* All patients who have benefited from an Implantable Loop recorder in the Nancy's Teaching Hospital

Exclusion Criteria:

* No Exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have benefited from an Implantable Loop recorder in the Nancy's Teaching Hospital between 1 January 2010 and 31 decembre 2019
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
significant bradycardia whitch result with an Indication of pacemaker implantation | At the moment of enregistrement of a significative arrhythmia or at the end of the 3 years of follow up
  2° and 3° AV block, sinus node dysfunction with pause > 8 sec or > 3sec with concomitant symptoms, sick sinus syndrom

SECONDARY OUTCOMES:
Patient group without benefit of implantation of the Implantable Loop Recorder | At the end of the 3 years of follow-up
  non significant bradicardia or arythmias revealed by loop recorder during monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- De Ciancio, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
anonymous individual datas for baseling pre implantatory caracteristcs and clinical outecome would be available
Supporting Information: SAP, ICF, CSR
Time Frame: 6 month
Access Criteria: Data access request will be reviewed by investigator team. Requestors will be required to signe a data access agreement

REFERENCES:
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Background] Edvardsson N, Wolff C, Tsintzos S, Rieger G, Linker NJ. Costs of unstructured investigation of unexplained syncope: insights from a micro-costing analysis of the observational PICTURE registry. Europace. 2015 Jul;17(7):1141-8. doi: 10.1093/europace/euu412. Epub 2015 Mar 10. PMID 25759408
- [Background] Padmanabhan D, Kancharla K, El-Harasis MA, Isath A, Makkar N, Noseworthy PA, Friedman PA, Cha YM, Kapa S. Diagnostic and therapeutic value of implantable loop recorder: A tertiary care center experience. Pacing Clin Electrophysiol. 2019 Jan;42(1):38-45. doi: 10.1111/pace.13533. Epub 2018 Dec 4. PMID 30357866